CLINICAL TRIAL: NCT07243288
Title: Evaluation of an Early Radiomic Signature in Patients With Metastatic Pancreatic Adenocarcinoma Treated With First-line Chemotherapy
Acronym: RADIOPAN
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: DAT23014
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer; MeSH Term-Pancreatic Cancer, Adult)
Keywords: Pancreatic cancer; Radiomics; RWE epidemiology; Prognosis prediction
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Folfox protocol; folfirinox; Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADK: All adult patients diagnosed with pancreatic cancer at AP-HP hospitals, identified using ICD-10 codes (C25)
  Interventions: Drug: Patients treated with FOLFOX or FOLFIRINOX in first line; Drug: Patients treated with GEMCITABINE in first line

INTERVENTIONS:
Drug: Patients treated with FOLFOX or FOLFIRINOX in first line — Treatment with FOLFOX or FOLFIRINOX (chemotherapy protocols) in first line
Drug: Patients treated with GEMCITABINE in first line — Treatment with GEMCITABINE (chemotherapy protocols) in first line

SUMMARY:
Pancreatic cancer, which has a poor prognosis, is becoming increasingly common in industrialized countries. Chemotherapy is the main treatment available for metastatic disease. Response to chemotherapy is currently assessed using imaging to monitor changes in the size of lesions undergoing treatment. Radiomics is a new method of analyzing quantitative data extracted from imaging that can be used to develop prediction algorithms and evaluate response to treatment. There is little robust radiomics data available for evaluating response to first-line treatments for pancreatic adenocarcinoma. Our main hypothesis is that quantifying tumor-related architectural changes could enable early identification of patients who will not respond to chemotherapy.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma is a cancer with a poor prognosis, and its incidence is increasing, particularly in industrialized countries. Systemic chemotherapy, the main treatment available, has improved survival in patients with metastatic pancreatic adenocarcinoma. Following the results of the study by Conroy et al., the combination of 5FU + oxaliplatin + irinotecan (FOLFIRINOX) is one of the standard first-line chemotherapy regimens for metastatic pancreatic adenocarcinoma.

The population of patients with metastatic pancreatic adenocarcinoma is heterogeneous, with different survival profiles. This is part of a multifactorial picture that is still poorly understood (molecular, terrain, other factors, etc.). Response to chemotherapy is currently assessed using the RECIST 1.1 method, which takes into account changes in the size of lesions during treatment. However, this method is sometimes limited, as it does not always take into account the underlying pathophysiology.

Radiomics consists of analyzing quantitative data extracted from imaging, which allows prediction algorithms to be developed. Several studies have suggested that tumor architecture could be a biomarker of response and survival in patients with esophageal, lung, or colorectal cancer.

A study of 41 patients with advanced pancreatic cancer treated with gemcitabine-based chemotherapy evaluated the impact of radiological architectural assessment on treatment response. The results showed that tumor size, asymmetry, and standard deviation of density at baseline were associated with progression-free survival, and that tumor size and standard deviation of density at baseline were associated with overall survival. These results remain to be confirmed in a larger population, hence the value of conducting our work with data from our database.

Our main hypothesis is that quantifying tumor-related architectural changes could enable early identification of patients who will not respond to treatment. The overall objective would be to tailor the therapeutic strategy to each individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Diagnosis of acute alcoholic hepatitis (ICD10 C25) in a pathology report, followed by manual verification in clinical documents

Exclusion Criteria:

* Patients younger than 18 years at diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pancreatic cancer across all AP-HP hospitals. Data will be collected retrospectively from the AP-HP Clinical Data Warehouse (EDS).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival after diagnosis of pancreatic cancer | From diagnosis up to 7 years after
  Overall survival will be assessed using mortality data recorded in the AP-HP Clinical Data Warehouse. The objective is to evaluate prognosis and identify risk factors associated with death after a diagnosis of pancreatic cancer, by integrating clinical, biological, histological and radiomics information. Survival will be analysed at multiple time points, including 1 month, 6 months, and 1 year after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Anna PELLAT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Bartoli M, Barat M, Dohan A, Gaujoux S, Coriat R, Hoeffel C, Cassinotto C, Chassagnon G, Soyer P. CT and MRI of pancreatic tumors: an update in the era of radiomics. Jpn J Radiol. 2020 Dec;38(12):1111-1124. doi: 10.1007/s11604-020-01057-6. Epub 2020 Oct 21. PMID 33085029
- [Background] Cheng SH, Cheng YJ, Jin ZY, Xue HD. Unresectable pancreatic ductal adenocarcinoma: Role of CT quantitative imaging biomarkers for predicting outcomes of patients treated with chemotherapy. Eur J Radiol. 2019 Apr;113:188-197. doi: 10.1016/j.ejrad.2019.02.009. Epub 2019 Feb 11. PMID 30927946